CLINICAL TRIAL: NCT00687973
Title: Effect of the Fixed Dose Combination Amlodipine/Valsartan on Central Aortic Blood Pressure in Uncontrolled Essential Hypertension With Amlodipine 5 mg
Acronym: EXPLOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489AFR02
Record Dates: First submitted 2008-03-20; First posted 2008-06-02 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valsartan/amlodipine 160/10 mg (Experimental): Patients were treated with valsartan/amlodipine 80/5 mg for 8 weeks followed by forced uptitration to valsartan/amlodipine 160/10 mg for 16 weeks. All doses were taken orally once daily in the morning, except on days when clinic visits were scheduled.
  Interventions: Drug: Valsartan/amlodipine 80/5 mg tablets
- Atenolol/amlodipine 100/10 mg (Active Comparator): Patients were treated with atenolol/amlodipine 50/5 mg for 8 weeks followed by forced uptitration to atenolol/amlodipine 100/10 mg for 16 weeks. All doses were taken orally once daily in the morning, except on days when clinic visits were scheduled.
  Interventions: Drug: Amlodipine 5 mg capsules; Drug: Amlodipine 10 mg capsules; Drug: Atenolol 50 mg tablets; Drug: Atenolol 100 mg tablets

INTERVENTIONS:
Drug: Valsartan/amlodipine 80/5 mg tablets
  Arms: Valsartan/amlodipine 160/10 mg
Drug: Amlodipine 5 mg capsules
  Arms: Atenolol/amlodipine 100/10 mg
Drug: Amlodipine 10 mg capsules
  Arms: Atenolol/amlodipine 100/10 mg
Drug: Atenolol 50 mg tablets
  Arms: Atenolol/amlodipine 100/10 mg
Drug: Atenolol 100 mg tablets
  Arms: Atenolol/amlodipine 100/10 mg

SUMMARY:
Assess that for an equivalent brachial blood pressure (BP)lowering, a fixed dose combination amlodipine/valsartan based regimen reduces central aortic BP pressure to a larger extent than an atenolol/amlodipine combination based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Hypertension defined by MSDBP > 90 and or MSSBP > 140 mmHg, MSDBP > 80 mmHg, or/and MSSBP > 130 mmHg if diabetes or chronic renal impairment uncontrolled under their previous therapy, or untreated , or experiencing unacceptable side effects
* Written informed consent to participate in the study prior to any study procedures

Exclusion Criteria:

* Severe hypertension (grade 3 WHO classification MSDBP > 110 mmHg and/or MSSBP > 180 mmHg)
* Evidence of a secondary form of hypertension
* Type 1 diabetes mellitus
* History of congestive heart failure, unstable coronary insufficiency, life threatening arrhythmia, significant valvular disease, second or third degree heart block etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- 2 & 4 rue Lionel Terray BP 308, Rueil-Malmaison, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Started | 193 | 200
Completed | 169 | 162
Not Completed | 24 | 38
Not completed — Adverse Event | 18 | 28
Not completed — Lack of Efficacy | 2 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Administrative Reasons | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg | Total
Number analyzed (Participants) | 193 | 200 | 393
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.94) | 56.2 (11.09) | 56.9 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 101 | 183
  Male | 111 | 99 | 210
Region of Enrollment [Number; unit: participants]
  France | 193 | 200 | 393

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Central Systolic Blood Pressure (SBP) at Week 24 (Radial Measurement)
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 176 | 178
mmHg | -13.65 (1.15) | -9.7 (1.09)

2. Secondary Outcome: Change From Baseline of Central Systolic Blood Pressure (SBP) at Week 8 (Radial Measurement)
Time Frame: Baseline and Week 8
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 183 | 189
mmHg | -10.92 (1.18) | -8.3 (1.12)

3. Secondary Outcome: Change From Baseline of Central Pulse Pressure at Week 24 (Radial Measurement)
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 176 | 178
mmHg | -5.5 (0.65) | -1.7 (0.63)

4. Secondary Outcome: Change From Baseline of Augmentation Index (Aix) at Week 8
Description: To calculate the blood pressure augmentation index, the inflection point of the pressure curve corresponding to the return of the reflection wave was determined. The ratio between the pressure located above and below the inflection point was calculated.
Time Frame: Baseline and Week 8
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 181 | 187
Ratio | -2.21 (0.78) | 3.61 (0.76)

5. Secondary Outcome: Change From Baseline of Aix at Week 24
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 175 | 178
Ratio | -4.10 (0.72) | 2.40 (0.70)

6. Secondary Outcome: Change From Baseline of Aix Corrected to Heart Rate at Week 24
Description: The heart rate correction was computed by a multivariate model analysis
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 169 | 170
Ratio | -4.12 (0.67) | -2.43 (0.66)

7. Secondary Outcome: Change From Baseline of Pulse Wave Velocity at Week 24 (Radial Measurement)
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population; Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 139 | 147
m/s | -0.98 (0.18) | -0.95 (0.17)

8. Secondary Outcome: Change From Baseline of Brachial SBP/DBP at Week 24 (Tonometry Center)
Description: Applanation tonometry is a measurement of aortic pressure and vascular stiffness. To assess the central aortic blood pressure, it is necessary to calibrate the applanation tonometry device using the brachial blood pressure.
Time Frame: Baseline and Week 24
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 176 | 176
mmHg
  SBP | -12.93 (1.14) | -11.78 (1.11)
  DBP | -7.85 (0.70) | -7.94 (0.68)

9. Secondary Outcome: Change From Baseline of Brachial Pulse Pressure at Week 24 (Tonometry Center)
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 176 | 176
mmHg | -5.02 (0.72) | -3.66 (0.70)

10. Secondary Outcome: Change From Baseline of SBP/DBP at Week 24 (Office BP)
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 183 | 185
mmHg
  SBP | -14.49 (1.08) | -16.94 (1.07)
  DBP | -8.17 (0.72) | -10.45 (0.71)

11. Secondary Outcome: Change From Baseline of Pulse Pressure at Week 24 (Office BP)
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Number analyzed (Participants) | 183 | 185
mmHg | -6.32 (0.81) | -6.48 (0.81)

ADVERSE EVENTS:
Groups:
- Amlodipine 5 mg: Run-in: Amlodipine 5 mg
Arm/Group | Amlodipine 5 mg | Valsartan/Amlodipine 160/10 mg | Atenolol/Amlodipine 100/10 mg
Serious Adverse Events (participants affected / at risk) | 3/393 | 4/193 | 4/200
Other Adverse Events (participants affected / at risk) | 10/393 | 30/193 | 31/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5 mg (N=393) | Valsartan/Amlodipine 160/10 mg (N=193) | Atenolol/Amlodipine 100/10 mg (N=200)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 0 | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Joint arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5 mg (N=393) | Valsartan/Amlodipine 160/10 mg (N=193) | Atenolol/Amlodipine 100/10 mg (N=200)
Oedema peripheral (General disorders) | 10 | 30 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However,Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.